CLINICAL TRIAL: NCT00003711
Title: A Phase I Trial of LY231514 With Irinotecan Administered Intravenously Every 21 Days in Patients With Metastatic Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: San Antonio Cancer Institute (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: LILLY-H3E-MC-JMAX(a); UTHSC-9675011396; CDR0000066819 (Registry Identifier: PDQ (Physician Data Query)); SACI-IDD-97-08; NCI-V98-1505
Record Dates: First submitted 1999-11-01; First posted 2004-09-14 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2000-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Irinotecan; Pemetrexed

INTERVENTIONS:
Drug: irinotecan hydrochloride
Drug: pemetrexed disodium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy with pemetrexed disodium and irinotecan in treating patients who have metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of LY231514 followed by irinotecan in patients with metastatic cancer. II. Determine the quantitative and qualitative toxicity of LY231514 in combination with irinotecan in these patients. III. Assess plasma pharmacokinetics in these patients treated with this regimen. IV. Document any antitumor activity of this regimen in these patients.

OUTLINE: This is a dose escalation study. Patients receive LY231514 IV over 10 minutes followed by irinotecan IV over 90 minutes on day 1. Courses repeat every 3 weeks in the absence of disease progression and unacceptable toxicity. Cohorts of 3-6 patients each receive escalating doses of LY231514 and irinotecan. If escalation of one drug in the combination results in unacceptable dose limiting toxicity (DLT), the drug is not escalated further. Instead, the dose of that drug is decreased to its safe dose, and the second drug is escalated until unacceptable DLT results. If DLT occurs in 2 of up to 6 patients at any level, dose escalation is stopped. The maximum tolerated dose is defined as the highest dose at which fewer than 2 of 6 patients experience DLT during courses 1 or 2.

PROJECTED ACCRUAL: Up to 42 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven metastatic solid tumors that are refractory to standard therapies or for which no potentially effective therapy exists No leukemia, lymphoma, or multiple myeloma Measurable or evaluable disease No pleural or peritoneal effusions No symptomatic brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute granulocyte count at least 1500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9.0 g/dL Hepatic: Bilirubin normal AST and ALT no greater than 3 times normal (no greater than 5 times normal if liver involvement present) Albumin at least 2.5 g/dL Renal: Creatinine clearance at least 45 mL/min Other: Not pregnant or nursing Fertile patients must use effective contraception during and for 3 months after study No active infection No concurrent serious systemic disorders Body surface area no greater than 3.0 m2

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Chemotherapy: At least 3 weeks since prior chemotherapy and recovered No prior LY231514 or irinotecan No greater than 6 prior courses of a regimen containing an alkylating agent (except low dose cisplatin) No greater than 4 prior courses of a carboplatin-containing regimen No prior mitomycin No other concurrent chemotherapy Endocrine therapy: No concurrent hormone therapy (except contraceptives or corticosteroids) Radiotherapy: No prior radiotherapy to 25% or more of the bone marrow No prior radiotherapy to the whole pelvis Recovered from any prior radiotherapy No concurrent radiotherapy Surgery: Not specified Other: At least 4 weeks since any prior investigational agents No concurrent experimental medications No aspirin or other nonsteroidal antiinflammatory agents for 2 days prior, the day of, and 2 days after the dose of LY231514 (5 days prior to LY231514 for long acting agents such as piroxicam)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-09; Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Johnson, MD, Study Chair — San Antonio Cancer Institute
Locations (2):
- United States (2):
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - San Antonio Cancer Institute, San Antonio, Texas